CLINICAL TRIAL: NCT00764179
Title: Effects (Long Term Analysis) of an Hyperproteinic Nutrition on Neonates With Intra-uterine Growth Delay : a Prospective, Multicentric , Randomized, Double Blind Study ("Proneonat")
Acronym: Proneonat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of recruitment, high number of patients lost to follow-up
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRD/06/12-P
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Intra-uterine Growth Delay
Keywords: Neonates with intra-uterine growth delay
MeSH Terms: interventions — Proteins; Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): hyperproteinic milk
  Interventions: Other: milk enriched in proteins (2.15 g/100ml)
- 2 (Active Comparator): Normoproteinic milk
  Interventions: Other: milk with normal protein concentration (1.45g/100ml)

INTERVENTIONS:
Other: milk enriched in proteins (2.15 g/100ml) — Neonates will drink the hyperproteinic milk until they reach the 25th of "Sempé and Pedron" curve (milk to be taken at least until 40 weeks of amenorrhoea or at maximum until 4 months of corrected age)
  Arms: 1
Other: milk with normal protein concentration (1.45g/100ml) — Neonates will drink the normoproteinic milk until they reach the 25th of "Sempé and Pedron" curve (milk to be taken at least until 40 weeks of amenorrhoea or at maximum until 4 months of corrected age)
  Arms: 2

SUMMARY:
Neonates with intra-uterine growth delay represent more than 2% of the 800 000 annual births in France. Studies have shown that milks enriched with protein allow to accelerate newborns growth. According to some papers, growth acceleration would have a favourable effect on psycho-motor development at age of 2 or 3. However, for other authors, this would not lead to any benefit and even an early hyperproteinic feeding would have bad long term consequences such as appearance of several diseases in the future adult (overweight, diabetes, arterial hypertension, renal function alteration).The main objective of this clinical trial is to check that an hyperproteinic feeding does not lead to any benefit on psycho-motor development at age of 2, compared with a milk containing same level of protein than milk proposed to newborns of normal weight. The secondary objectives of our clinical trial are to compare the effects of these two types of milk on renal function, arterial blood pressure, body composition, corpulence, food preferences, insulin resistance and intestinal integrity at age of 2. A sub study will also be realized to analyse the proteic turn over . This sub-study will be undertaken only with neonates of Nantes Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with intra-uterine growth delay (with weight < 10th centile)
* Aged >34 weeks of amenorrhoea
* For neonates >38 weeks of amenorrhoea, weight < 2500g
* Mother's refusal of breast feeding
* Informed consent signed by the 2 parents
* Possibility to follow newborns until age of 2

Exclusion Criteria:

* Subject not fulfilling inclusion criteria
* Severe disease (syndrome and/or congenital abnormality, deficiency of metabolism at birth)

Ages: 34 Weeks to 39 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2008-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quotient of psycho-motor development evaluated by the Brunet-Lezine test at age of 2 | at 2 years old

SECONDARY OUTCOMES:
Leptine, glycemia/insulin and pro-insulin blood level | At age of 15 (+/- 2) days and at age of 2 years
Plasmatic and urinary citrulline levels | At age of 15 (+/- 2) days and at age of 2 years
Micro-albuminuria, creatinine, urea, sodium and potassium urine levels | At age of 15 (+/- 2) days and at age of 2 years
Faecal floa, faecal calprotectine and other markers | At age of 15 (+/- 2) days and at age of 2 years
Arterial blood pressure, arterial elasticity, adiponectine, preferential food choices, kidney size | at age of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DARMAUN, Professor, Study Director — Nantes Universitary Hospital; Dominique DARMAUN, Professor, Principal Investigator — Nantes Universitary Hospital; Jean-Christophe ROZE, Professor, Study Chair — Nantes Universitary Hospital; Clotilde DES ROBERT, Doctor, Study Chair — Nantes Universitary Hospital; Umberto SIMEONI, Professor, Study Chair — AP-HM, "Hôpital de la conception- Marseille"; Régis HANKARD, Professor, Study Chair — CHU of Poitiers; Eric DUMAS DE LA ROQUE, Doctor, Study Chair — CHU of Bordeaux (Pellegrin-Tripode Hospital); Olivier BAUD, Professor, Study Chair — AP-HP (Paris - Robert Debré Hospital)
Locations (1):
- Universitary Hospital, Nantes, France